CLINICAL TRIAL: NCT04051541
Title: Simulation of Adenosine Push Methods for Treatment of SVT Using Agitated Saline Visualized by Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A18-400
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2019-08

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Intervention Model Description: This is a simulation study in which all participants receive a dose of agitated saline through an IV using three different administration methods.
Masking Description: The investigator performing the ultrasound and the person timing the simulation were both blind to the method used for each push. An unblended investigator performed the pushes but did not assess the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulation arm (Other): All patients were entered into the Simulation arm and received 3 pushes of agitated saline via 3 different methods of delivery. All patients received all methods. The order of the methods for each patient was randomized.
  Interventions: Other: Agitated saline push

INTERVENTIONS:
Other: Agitated saline push — Push of agitated saline to simulate adenosine used for supraventricular tachycardia

SUMMARY:
Supraventricular tachycardia (SVT) is an abnormally fast heart rhythm arising from improper electrical activity in the upper part of the heart. SVT is commonly treated with adenosine using three different IV administration techniques. However, it is not well known which of these three techniques is the quickest or most likely to reach the heart in order to stop SVT. This study will simulate each of those techniques in an investigator-blinded procedure. Intravenous agitated saline, used as a surrogate for a dose of adenosine, will be administered to healthy volunteers using all three techniques and monitored using bedside ultrasound to observe their efficacy and speed in reaching the right side of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18 years and older
* Able to understand and provide signed consent for the study
* Must be healthy; not being actively treated for any condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being, as evaluated by study investigator

Exclusion Criteria:

* Non-English speaker
* Those with contraindications to peripheral IV placement, such as infection or other contraindication noted from evaluation by study investigator
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Time to ultrasound visualization of agitated saline in the right heart | <5 seconds
  Time from IV push to ultrasound visualization of agitated saline in the right heart

CONTACTS AND LOCATIONS:
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murman DH, McDonald AJ, Pelletier AJ, Camargo CA Jr. U.S. emergency department visits for supraventricular tachycardia, 1993-2003. Acad Emerg Med. 2007 Jun;14(6):578-81. doi: 10.1197/j.aem.2007.01.013. Epub 2007 Apr 20. PMID 17449792
- [Background] Brubaker S, Long B, Koyfman A. Alternative Treatment Options for Atrioventricular-Nodal-Reentry Tachycardia: An Emergency Medicine Review. J Emerg Med. 2018 Feb;54(2):198-206. doi: 10.1016/j.jemermed.2017.10.003. Epub 2017 Nov 26. PMID 29239759
- [Background] Alabed S, Sabouni A, Providencia R, Atallah E, Qintar M, Chico TJ. Adenosine versus intravenous calcium channel antagonists for supraventricular tachycardia. Cochrane Database Syst Rev. 2017 Oct 12;10(10):CD005154. doi: 10.1002/14651858.CD005154.pub4. PMID 29025197
- [Background] Weberding NT, Saladino RA, Minnigh MB, Oberly PJ, Tudorascu DL, Poloyac SM, Manole MD. Adenosine Administration With a Stopcock Technique Delivers Lower-Than-Intended Drug Doses. Ann Emerg Med. 2018 Feb;71(2):220-224. doi: 10.1016/j.annemergmed.2017.09.002. Epub 2017 Oct 28. PMID 29089171
- [Background] Losek JD, Endom E, Dietrich A, Stewart G, Zempsky W, Smith K. Adenosine and pediatric supraventricular tachycardia in the emergency department: multicenter study and review. Ann Emerg Med. 1999 Feb;33(2):185-91. doi: 10.1016/s0196-0644(99)70392-6. PMID 9922414
- [Background] Kleinman ME, Chameides L, Schexnayder SM, Samson RA, Hazinski MF, Atkins DL, Berg MD, de Caen AR, Fink EL, Freid EB, Hickey RW, Marino BS, Nadkarni VM, Proctor LT, Qureshi FA, Sartorelli K, Topjian A, van der Jagt EW, Zaritsky AL. Part 14: pediatric advanced life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S876-908. doi: 10.1161/CIRCULATIONAHA.110.971101. No abstract available. PMID 20956230
- [Background] Madsen CD, Pointer JE, Lynch TG. A comparison of adenosine and verapamil for the treatment of supraventricular tachycardia in the prehospital setting. Ann Emerg Med. 1995 May;25(5):649-55. doi: 10.1016/s0196-0644(95)70179-6. PMID 7741343
- [Background] Neumar RW, Otto CW, Link MS, Kronick SL, Shuster M, Callaway CW, Kudenchuk PJ, Ornato JP, McNally B, Silvers SM, Passman RS, White RD, Hess EP, Tang W, Davis D, Sinz E, Morrison LJ. Part 8: adult advanced cardiovascular life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S729-67. doi: 10.1161/CIRCULATIONAHA.110.970988. PMID 20956224
- [Background] Ng GA, Martin W, Rankin AC. Imaging of adenosine bolus transit following intravenous administration: insights into antiarrhythmic efficacy. Heart. 1999 Aug;82(2):163-9. doi: 10.1136/hrt.82.2.163. PMID 10409529
- [Background] Wen M, Stock K, Heemann U, Aussieker M, Kuchle C. Agitated saline bubble-enhanced transthoracic echocardiography: a novel method to visualize the position of central venous catheter. Crit Care Med. 2014 Mar;42(3):e231-3. doi: 10.1097/CCM.0000000000000130. PMID 24317496
- [Background] Duran-Gehring PE, Guirgis FW, McKee KC, Goggans S, Tran H, Kalynych CJ, Wears RL. The bubble study: ultrasound confirmation of central venous catheter placement. Am J Emerg Med. 2015 Mar;33(3):315-9. doi: 10.1016/j.ajem.2014.10.010. Epub 2014 Oct 13. PMID 25550065
- [Background] Gekle R, Dubensky L, Haddad S, Bramante R, Cirilli A, Catlin T, Patel G, D'Amore J, Slesinger TL, Raio C, Modayil V, Nelson M. Saline Flush Test: Can Bedside Sonography Replace Conventional Radiography for Confirmation of Above-the-Diaphragm Central Venous Catheter Placement? J Ultrasound Med. 2015 Jul;34(7):1295-9. doi: 10.7863/ultra.34.7.1295. PMID 26112633
- [Background] Weekes AJ, Johnson DA, Keller SM, Efune B, Carey C, Rozario NL, Norton HJ. Central vascular catheter placement evaluation using saline flush and bedside echocardiography. Acad Emerg Med. 2014 Jan;21(1):65-72. doi: 10.1111/acem.12283. PMID 24552526
- [Background] Ketkar VA, Kolling WM, Nardviriyakul N, VanDer Kamp K, Wurster DE. Stability of undiluted and diluted adenosine at three temperatures in syringes and bags. Am J Health Syst Pharm. 1998 Mar 1;55(5):466-70. doi: 10.1093/ajhp/55.5.466. PMID 9522931
- [Background] Green AP, Giattina KH. Adenosine administration for neonatal SVT. Neonatal Netw. 1993 Aug;12(5):15-8. PMID 8350844